CLINICAL TRIAL: NCT01782989
Title: A Randomized, Double Blind, Placebo Controlled Study Evaluating ORACEA® in Subjects With Geographic Atrophy Secondary to Non-Exudative Age-Related Macular Degeneration
Brief Title: Clinical Study to Evaluate Treatment With ORACEA® for Geographic Atrophy (TOGA)
Acronym: TOGA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Paul Yates, MD, PhD (Other)
Collaborators: MEDARVA Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Paul Yates, MD, PhD, Associate Professor of Ophthalmology, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16586
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Geographic Atrophy
Keywords: geographic atrophy; non-exudative age-related macular degeneration; macular degeneration; dry macular degeneration; dry AMD
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ORACEA® (Experimental): 40mg doxycycline
  Interventions: Drug: ORACEA®
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ORACEA® — ORACEA® (40mg doxycycline) capsule daily for 24 months
  Arms: ORACEA®
Drug: Placebo — Placebo capsule daily for 24 months
  Arms: Placebo

SUMMARY:
This is a prospective, randomized study to evaluate the efficacy and safety of ORACEA® in the treatment of geographic atrophy due to dry age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
Eligible participants will complete a 6-month Observation Phase, followed by a 24-month Treatment Phase, followed by an End of Study Visit. Eligible participants will be randomized at Month 6 in a 1:1 ratio to either ORACEA (40 mg doxycycline) or placebo capsule to be taken once-daily for 24 months. Over the course of the 31-month study, a total of 9 clinic visits and 3 telephone calls are required.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age >/=55 years
* Best corrected visual acuity of 20/20 - 20/400 in the study eye
* Best corrected visual acuity of hand motion or better in the non-study eye
* Clinical diagnosis of geographic atrophy secondary to non-exudative age-related macular degeneration in at least one eye (study eye)
* Geographic atrophy lesions of ≥ 0.5 and ≤ 7.0 MPS disc areas

Exclusion Criteria:

* History of or active presence of choroidal neovascularization secondary to exudative age-related macular degeneration in the study eye
* History of or active presence of choroidal neovascularization secondary to exudative age-related macular degeneration in the non-study eye requiring any treatment within 12 months prior to Day 0 or expected to require treatment for the duration of the study
* Prior treatment for non-exudative age-related macular degeneration
* Current or previous history of treatment of the study eye with any tetracycline derivative for any ocular condition.
* History of vitreoretinal surgery, corneal transplant, or laser photocoagulation in the study eye
* Any intraocular or periocular surgery within 90 days prior to Day 0 in the study eye.
* History of any hypersensitivity to tetracycline components
* Use of a tetracycline derivative therapy for a concurrent systemic or ocular disorder within 90 days of Day 0
* History of sensitivity to the sun

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2013-02; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Rate of enlargement in area of geographic atrophy in the study eye during the treatment period. | Month 6 and Month 30

SECONDARY OUTCOMES:
Change in Best Corrected Visual Acuity (BCVA) | Month 6 and Month 30

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Yates, MD, PhD, Principal Investigator — University of Virginia
Locations (37):
- United States (37):
  - Macula and Retina Institute, Glendale, California
  - Retina Consultants of San Diego, Poway, California
  - Colorado Retina Associates, PC, Golden, Colorado
  - Eldorado Retina Associates, Louisville, Colorado
  - New England Retina Associates, Hamden, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Medical Center Eye Institute / Gulf Region Clinical Research Institute, Pensacola, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Gailey Eye Clinic, Bloomington, Illinois
  - Retina Associates of Kentucky, Lexington, Kentucky
  - New England Eye Center at Tufts Medical Center, Boston, Massachusetts
  - Harvard Vanguard Medical Associates, Boston, Massachusetts
  - Vitreo-Retinal Associates, Worcester, Massachusetts
  - Retina Specialists of Michigan, Grand Rapids, Michigan
  - Retina Center, Minneapolis, Minnesota
  - Lifelong Vision Foundation, Chesterfield, Missouri
  - Delaware Valley Retina Associates, Lawrenceville, New Jersey
  - Retinal and Ophthalmic Consultants, Northfield, New Jersey
  - New Jersey Retina, Toms River, New Jersey
  - MaculaCare, New York, New York
  - Vitreous Retina Macula Consultants of New York, New York, New York
  - New York Eye and Ear, New York, New York
  - Retina Associates of Western New York, Rochester, New York
  - Cole Eye Institute / Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Retina, Eugene, Oregon
  - Pennsylvania Retina Specialists, PC, Camp Hill, Pennsylvania
  - Mid Atlantic Retina / Wills Eye Institute, Philadelphia, Pennsylvania
  - University of Pittsburgh Eye Center, Pittsburgh, Pennsylvania
  - Associates in Ophthalmology, Ltd, West Mifflin, Pennsylvania
  - Retina Research Institute of Texas, Abilene, Texas
  - Brian B. Berger, MD and Associates / Retina Research Center, Austin, Texas
  - Retina Associates of South Texas, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Wagner Macula & Retina Center, Virginia Beach, Virginia
  - Virginia Retina Center, Warrenton, Virginia
  - Retina Cosultants, Charleston, West Virginia

REFERENCES:
- [Derived] Dalvi S, Roll M, Chatterjee A, Kumar LK, Bhogavalli A, Foley N, Arduino C, Spencer W, Reuben-Thomas C, Ortolan D, Pebay A, Bharti K, Anand-Apte B, Singh R. Human iPSC-based disease modeling studies identify a common mechanistic defect and potential therapies for AMD and related macular dystrophies. Dev Cell. 2024 Dec 16;59(24):3290-3305.e9. doi: 10.1016/j.devcel.2024.09.006. Epub 2024 Oct 2. PMID 39362220